CLINICAL TRIAL: NCT00851591
Title: Effect of Fenugreek on Milk Production
Acronym: fenugreek
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment; investigator chose not to continue study
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A08-3479
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Lactation
Keywords: fenugreek; galactogogue; breastmilk; Trigonella foenum-graecum; Bird's Foot; Greek Clover; Greek Hay; Hu Lu Ba; Trigonella
MeSH Terms: conditions — Breast Feeding | interventions — fenugreek seed meal; Psyllium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fenugreek category 1 (Experimental): receive fenugreek
  Interventions: Drug: fenugreek
- Placebo Category 2 (Placebo Comparator): receive placebo
  Interventions: Drug: Placebo (Psyllium)

INTERVENTIONS:
Drug: fenugreek — 3 capsules 3 times per day with a full glass of water each dose for 7 days
  Other Names: Trigonella foenum-graecum, Alhova, Bird's Foot, Greek Clover
  Arms: Fenugreek category 1
Drug: Placebo (Psyllium) — 3 capsules 3 times a day with a full glass of water each dose for 7 days
  Other Names: Metamucil®,; Hydrocil Instant®,; Modane Bulk Powder®
  Arms: Placebo Category 2

SUMMARY:
Each year, approximately 3 million mothers in the USA alone leave the hospital breastfeeding an infant. However, a large number discontinue breastfeeding, because milk synthesis is poor or simply stops. Termed "Insufficient Milk Syndrome," this condition probably accounts for approximately 5-10% of the total population of breastfeeding mothers and includes many mothers with premature infants, mothers with polycystic ovary syndrome, and a myriad of other unknown causes. The mother's inability to breastfeed causes enormous feelings of inadequacy, grief, depression, and other problems, not to mention increased health risks to the infant.

The most popular herbal remedy used around the world for increasing milk synthesis is fenugreek. Fenugreek (Trigonella foenum graecum) is a seed product from the legume family that is commonly sold, since the dried, ripe seed and extracts are used as an artificial flavor for maple syrup. When used orally in amounts commonly found in foods, it has been granted Generally Recognized as Safe (GRAS) status in the USA by the FDA. Although it is used by millions of women around the world to increase their milk supply, we have only one small case report which suggested it might actually increase the milk supply.

In this one study, the authors found an approximate 40% increase in milk production, although the study was not blinded, nor did they use a control population. For these reasons, we still do not know with certainty if fenugreek works as a galactagogue.

This study is designed to accurately determine if seven days of fenugreek will stimulate milk production in a selected group of subjects with poor milk supply. We hypothesize that the women enrolled in the test group will have increased milk production at the end of the 8-day study.

DETAILED DESCRIPTION:
This study is designed to accurately determine if seven days of fenugreek will stimulate milk production in a selected group of subjects with poor milk supply. We hypothesize that the women enrolled in the test group will have increased milk production at the end of the 8-day study.

ELIGIBILITY:
Inclusion Criteria:

* Mothers 2-12 weeks postpartum
* Mothers with term infants 37 weeks gestation or older
* Mothers with poor milk supply documented by professional lactation consultants
* Mothers whose milk supply is less than 600 cc per 24 hours
* Mothers who agree not to breastfeed or provide their milk to their infants during this study

Exclusion Criteria:

* Mothers with documented mastitis
* Mothers with breast engorgement
* Mothers with inverted nipples
* Maternal BMI greater than 35
* Mothers currently consuming Reglan, Domperidone or other drugs/herbals used to induce milk production
* Mothers who are clinically ill or hospitalized, or taking the following medications:

  1. Diuretics
  2. Pseudoephedrine
  3. Anticholinergics
  4. Warfarin or any anticoagulant
  5. An estrogen-containing birth control pill
* Mothers with Diabetes mellitus
* Mothers who have had breast surgery that could alter milk synthesis or production
* Mothers diagnosed with Polycystic ovary syndrome
* Mothers with tubular breasts or breasts with insufficient glandular tissue
* Mothers diagnosed with Asthma or atopic disease
* Mothers who are known to be allergic to peanuts or soybeans
* Mothers who are pregnant
* Mothers whose milk supply per 24 hours exceeds 600 mL
* Mothers with Obstetrical evaluation recommending exclusion

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2008-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Hale, PhD, Study Director — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas, United States

REFERENCES:
- [Derived] Foong SC, Tan ML, Foong WC, Marasco LA, Ho JJ, Ong JH. Oral galactagogues (natural therapies or drugs) for increasing breast milk production in mothers of non-hospitalised term infants. Cochrane Database Syst Rev. 2020 May 18;5(5):CD011505. doi: 10.1002/14651858.CD011505.pub2. PMID 32421208

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 patients were recruited to participate. Recruitment was stopped due to a similar study had already been published and the inability to recruit patients.
Groups:
- 1 Group Scheduled to Receive Fenugreek: fenugreek: 3 capsules 3 times per day with a full glass of water each dose for 7 days
- 2 Group Scheduled to Receive Placebo: Psyllium: 3 capsules 3 times a day with a full glass of water each dose for 7 days
Period: Overall Study
Arm/Group | 1 Group Scheduled to Receive Fenugreek | 2 Group Scheduled to Receive Placebo
Started | 2 (These 2 participants did not receive treatment.) | 1 (One received treatment.)
Completed | 0 | 1
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 Group Scheduled to Receive Placebo | 1 Group Scheduled to Receive Fenugreek | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Main Outcome Variable of This Study is the Quantity of Milk Produced.
Description: The single value of this variable was calculated average from day 0 and day 8.
Time Frame: "Day 0" , "Day 8"
Arm/Group | 2 Group Scheduled to Receive Placebo
Number analyzed (Participants) | 0

2. Secondary Outcome: Secondary Outcome Variables Are to Include Milk-fat Content and Protein Content.
Description: Milk-fat content was not measured in these samples as we had decided to close the study.
  Protein content was not measured in these samples as we had decided to close the study.
Time Frame: day 0; day 8
Population: 0 patient samples
Groups:
- Milk Fat and Milk Protein: Milk fat levels were not determined in these samples as we had already decided to close study.
  Milk Protein levels were not determined in these samples as we had already decided to close study.
Arm/Group | Milk Fat and Milk Protein
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- 1 Group Scheduled to Receive Fenugreek: Fenugreek Category: These patients were scheduled to take 3 capsules 3 times per day with a full glass of water and each dose was for 7 days.
- 2 Group Scheduled to Receive Placebo: Psyllium Category: These patients were scheduled to take 3 capsules 3 times a day with a full glass of water and each dose was for 7 days.
Arm/Group | 1 Group Scheduled to Receive Fenugreek | 2 Group Scheduled to Receive Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes